CLINICAL TRIAL: NCT02733081
Title: Simplified IUD Insertion Technique: A Randomized Controlled Trial
Brief Title: Simplified IUD Insertion Technique
Acronym: SIIT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul D Blumenthal, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-35138
Record Dates: First submitted 2016-02-09; First posted 2016-04-11 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Contraception
Keywords: Long Acting Reversible Contraception; Intrauterine Device (IUD); Intrauterine Device (IUD) Insertion; Family Planning; International Family Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Traditional IUD Insertion (No Intervention): Standard IUD insertion according to package insert. Bimanual pelvic exam to assess uterine size and position will be performed. Uterine sound will be used to measure depth of uterus prior to insertion.
- Arm 2: Simplified IUD Insertion (Experimental): Simplified, investigational IUD insertion performed. No bimanual pelvic exam or uterine sounding.
  Interventions: Procedure: Simplified IUD Insertion

INTERVENTIONS:
Procedure: Simplified IUD Insertion — IUD Insertion with no bimanual pelvic exam or uterine sounding.
  Arms: Arm 2: Simplified IUD Insertion

SUMMARY:
This is a randomized controlled trial that compares traditional IUD insertion with that of a no uterine sound, no bimanual pelvic exam approach. The investigators hypothesis is that IUD placement is safe and effective without pre-procedural assessment of uterine size, direction, or depth.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older presenting to contraceptive clinic in Gaborone, Botswana for IUD insertion and have ability to give informed consent.

Exclusion Criteria:

* Known contradictions to copper IUD, inability to comply with study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Correct IUD Placement Immediately Post-Insertion | Immediately post-insertion
  Percent of correct IUD placements between control (traditional IUD insertion) and experimental (simplified IUD insertion) groups at time of insertion as visualized by transvaginal ultrasound.

SECONDARY OUTCOMES:
Correct IUD Placements 4-6 Weeks Post-Insertion | 4-6 weeks post-insertion
  Percent of correct IUD placements between control (traditional IUD insertion) and experimental (simplified IUD insertion) groups at 4-6 weeks after insertion as visualized by transvaginal ultrasound.
Patient Satisfaction with IUD Insertion | Immediately Post-Insertion
  Visual Analogue Scale (VAS)
Patient Pain Scores (VAS) | Immediately Post-Insertion
  Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Blumenthal, MD, MPH, Principal Investigator — Stanford University

REFERENCES:
- [Background] Tayal VS, Crean CA, Norton HJ, Schulz CJ, Bacalis KN, Bliss S. Prospective comparative trial of endovaginal sonographic bimanual examination versus traditional digital bimanual examination in nonpregnant women with lower abdominal pain with regard to body mass index classification. J Ultrasound Med. 2008 Aug;27(8):1171-7. doi: 10.7863/jum.2008.27.8.1171. PMID 18645075
- [Background] Padilla LA, Radosevich DM, Milad MP. Limitations of the pelvic examination for evaluation of the female pelvic organs. Int J Gynaecol Obstet. 2005 Jan;88(1):84-8. doi: 10.1016/j.ijgo.2004.09.015. PMID 15617719
- [Background] Maguire K, Davis A, Rosario Tejeda L, Westhoff C. Intracervical lidocaine gel for intrauterine device insertion: a randomized controlled trial. Contraception. 2012 Sep;86(3):214-9. doi: 10.1016/j.contraception.2012.01.005. Epub 2012 Feb 9. PMID 22325115
- [Background] Canteiro R, Bahamondes MV, dos Santos Fernandes A, Espejo-Arce X, Marchi NM, Bahamondes L. Length of the endometrial cavity as measured by uterine sounding and ultrasonography in women of different parities. Contraception. 2010 Jun;81(6):515-9. doi: 10.1016/j.contraception.2010.01.006. Epub 2010 Mar 1. PMID 20472119
- [Background] Bahamondes MV, Monteiro I, Canteiro R, Fernandes Ados S, Bahamondes L. Length of the endometrial cavity and intrauterine contraceptive device expulsion. Int J Gynaecol Obstet. 2011 Apr;113(1):50-3. doi: 10.1016/j.ijgo.2010.10.013. Epub 2011 Jan 26. PMID 21272883
- [Background] Heinemann K, Reed S, Moehner S, Minh TD. Risk of uterine perforation with levonorgestrel-releasing and copper intrauterine devices in the European Active Surveillance Study on Intrauterine Devices. Contraception. 2015 Apr;91(4):274-9. doi: 10.1016/j.contraception.2015.01.007. Epub 2015 Jan 16. PMID 25601352
- [Background] Christensen K, et al. Simplifying Insertion of IUD Devices. Selected for poster presentation at FIGO 2015, Vancouver British Columbia.
- [Background] ESHRE Capri Workshop Group. Intrauterine devices and intrauterine systems. Hum Reprod Update. 2008 May-Jun;14(3):197-208. doi: 10.1093/humupd/dmn003. Epub 2008 Apr 9. PMID 18400840